CLINICAL TRIAL: NCT02484924
Title: The Risk of Major Bleeding With Novel Anti-platelets: A Comparison of Ticagrelor With Clopidogrel in a Real World Population of 5000 Patients Treated for Acute Coronary Syndrome
Acronym: ROBOT-ACS
Status: Completed | Type: Observational
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Collaborators: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other); Countess of Chester NHS Foundation Trust (Other); St Helens & Knowsley Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 680/15
Record Dates: First submitted 2015-06-26; First posted 2015-06-30 (Estimated); Last update posted 2022-06-09 (Actual); Status verified 2016-01

CONDITIONS: Acute Coronary Syndrome; Bleeding; Novel Anti-platelets; Ticagrelor; Clopidogrel
MeSH Terms: conditions — Acute Coronary Syndrome; Hemorrhage | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clopidogrel Group: Those patients treated with clopidogrel for ACS (before new guideline implementation)
- Ticagrelor Group: Those patients treated with ticagrelor for ACS (after new guideline implementation)
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Ticagrelor — No intervention- purely observational
  Other Names: Clopidogrel
  Groups: Ticagrelor Group

SUMMARY:
A retrospective real world analysis of bleeding events with ticagrelor compared to clopidogrel in ACS patients.

DETAILED DESCRIPTION:
Major bleeding after myocardial infarction portends a poor outcome. A balance is required between potency of platelet inhibition and risk of bleeding. Ticagrelor provides faster and more effective platelet inhibition than Clopidogrel. In the PLATO trial Ticagrelor reduced the incidence of cardiovascular death, myocardial infarction and stroke compared to Clopidogrel after ACS (acute coronary syndrome). Although there was no difference in overall bleeding there was more non-CABG related major bleeding with Ticagrelor. It has since been recommended, in addition to aspirin, in treatment of moderate-high risk ACS by both ESC (European Society of Cardiology) and NICE (National Institute for Clinical Excellence). There has been widespread adoption as first line therapy in UK hospitals. There remains potential concern about bleeding in a "real world" population compromising more high risk patients; particularly more elderly and female, than those in PLATO. The investigators intend to perform a large "real world" comparison of bleeding risk with Ticagrelor compared to Clopidogrel in a UK ACS population. The investigators plan an observational cohort study of patients presenting with ACS at 5 district general hospitals in Merseyside and Cheshire. The investigators will collect data retrospectively on 2500 patients treated with Clopidogrel prior to the guideline change and 2500 treated with Ticagrelor thereafter. The primary end point will be incidence of BARC 3-5 (Bleeding Academic Research Consortium) and PLATO major bleeding.

ELIGIBILITY:
Inclusion Criteria:

1. Patient commenced on clopidogrel for ACS prior to change of ACS guidelines, or tiacgrelor for same indication afterwards.

Exclusion Criteria:

1. Patient already taking the drug in question (clopidogrel or ticagrelor) prior to the ACS event
2. Patients under 18 years of age
3. Patients in whom the drug is stopped during the same hospital admission due to clinical judgement dictating that it is no longer indicated (this does not apply to patients in whom a bleeding event is the precipitant for stopping the drug)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All-comers treated for ACS above the age of 18 with either clopidogrel or ticagrelor
Sampling Method: Non-Probability Sample
Enrollment: 5225 (Actual)
Dates: Start 2010-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The incidence of major bleeding defined by both BARC (3-5) and PLATO definitions | 12 months from treatment starting
  bleeding event

SECONDARY OUTCOMES:
Incidence of minor bleeding as defined by BARC and PLATO | 12 months from treatment starting
  Minor bleeding
Incidence of gastrointestinal bleeding | 12 months from treatment starting
  GI bleeding
Incidence of intracranial bleeding | 12 months from treatment starting
  intracranial bleeding
Rate of major adverse cardiovascular events; myocardial infarction, stroke and cardiovascular death | 12 months from treatment starting
  MACE/ischaemic events
Mortality | 12 months from treatment starting
  all cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Aleem Khand, MBChB MRCP, Principal Investigator — University Hospital Aintree
Locations (1):
- University Hospital Aintree, Liverpool, United Kingdom

REFERENCES:
- [Derived] Mullen L, Stables R. Validation of HES coding for the detection of major bleeding events: insights from the ROBOT-ACS study. BMC Med Res Methodol. 2025 Feb 20;25(1):42. doi: 10.1186/s12874-025-02503-7. PMID 39979827
- [Derived] Mullen L, Meah MN, Elamin A, Aggarwal S, Shahzad A, Shaw M, Hasara J, Rashid M, Fisher M, Ali T, Patel B, Ding WY, Grainger R, Heseltine T, Kirmani BH, Obeidat M, Kasolo Y, Thatchil J, Khand A. Risk of Major Bleeding With Potent Antiplatelet Agents After an Acute Coronary Event: A Comparison of Ticagrelor and Clopidogrel in 5116 Consecutive Patients in Clinical Practice. J Am Heart Assoc. 2021 Apr 20;10(8):e019467. doi: 10.1161/JAHA.120.019467. Epub 2021 Apr 9. PMID 33834845